CLINICAL TRIAL: NCT02305745
Title: Determining the Risk Elevation After Maternity
Acronym: DREAM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Other Study IDs: 20140799-01H
Record Dates: First submitted 2014-11-28; First posted 2014-12-03 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preeclampsia- observational: 45 women with preeclampsia
  Interventions: Other: Observational
- No preeclampsia- observational: 10 women without preeclampsia
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational

SUMMARY:
Evaluating the long term cardiovascular risks of those mothers who have been diagnosed with preeclampsia in pregnancy.

DETAILED DESCRIPTION:
Preeclampsia is a complication of pregnancy that happens in about 5-7% of all births. It is diagnosed when a mother has high blood pressure in pregnancy combined with protein in the urine which is sign that the kidneys are not functioning properly. When a mother has preeclampsia, the placenta makes abnormal amounts of several important proteins that damage the lining of the mother's blood vessels. The blood vessel damage that occurs places women at up to 10 times higher risk of having a heart attack or stroke at a younger age than women who did not have preeclampsia. It usually takes between 8 and 15 years after preeclampsia is diagnosed for the first heart attack or stroke to occur.

Unfortunately, this blood vessel damage is usually silent, meaning that women and their doctors are not aware of it. This makes it hard to predict which women are at highest risk of a heart attack or stroke and therefore need extra medical care to prevent it. Abnormal levels of the placenta proteins in the blood (right after delivery and at three and six months after delivery) as well as abnormalities of the placenta itself may be the earliest way to predict which women with preeclampsia are at risk of premature heart disease or stroke.

The purpose of this study is to collect blood and placentas from women with preeclampsia and without preeclampsia to measure and compare the levels of proteins in the blood and find abnormalities of the placentas that are associated with preeclampsia. We will then see if these tests can predict which women will go on to develop high blood pressure and ultimately be at higher risk of premature heart attack or stroke after pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Women with a pregnancy complicated by pre-eclampsia and women who are healthy and have had a normal singleton pregnancy(controls)

Exclusion Criteria:

Women with any of the following conditions will be excluded in both the control & preeclampsia groups:

1. known kidney disease prior to pregnancy or laboratory evidence of proteinuria prior to pregnancy
2. diabetes (Type I, Type II or Gestational Diabetes)
3. known Cardiovascular Disease (myocardial infarction, angina, stroke, or transient ischemic attack
4. multiple pregnancies (twins or more)
5. who do not understand English or French will be excluded In addition to those listed above, for the control group, women must have no other major maternal pregnancy complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to enroll 40 participants in the study: 30 women who have been diagnosed with preeclampsia and 10 women who have had a normal pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Persistence of high blood pressure (hypertension) and cardiovascular biomarkers in the blood at 6 months after a pregnancy with preeclampsia | Six months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Dr Laura Gaudet, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided